CLINICAL TRIAL: NCT06978452
Title: Behavioural Development, Long-term Outcomes and Opportunities to Optimize Youth Mental Health Trajectories
Acronym: BLOOM
Status: Recruiting | Type: Observational
Sponsor: Douglas Mental Health University Institute (Other)
Responsible Party: Principal Investigator, Lena Palaniyappan, Principal Investigator, Douglas Mental Health University Institute
Other Study IDs: 2024-960
Record Dates: First submitted 2025-05-11; First posted 2025-05-18 (Actual); Last update posted 2025-05-18 (Actual); Status verified 2024-11

CONDITIONS: Depression - Major Depressive Disorder; Bipolar; Psychosis; Eating Disorder NOS; ADHD; Substance Use Disorder (SUD); OCD
Keywords: antecedents; mental health prevention; resilience; access to care; help-seeking; youth in needs; biomarker; speech; language; cognition
MeSH Terms: conditions — Psychotic Disorders; Feeding and Eating Disorders; Attention Deficit Disorder with Hyperactivity; Substance-Related Disorders; Speech; Language

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Biospecimen Retention: Samples With DNA — The Bloom study will collect from a sub-set of the participants a variety of biological samples. Venous blood will be collected for both plasma and serum, a dried blood spot card, and a saliva sample and buccal cells will be collected from swabbing their cheeks. Samples will either be sent for analysis or transformed into a derivative that will be analyzed. Serum samples will be analyzed for fasting glucose, insulin, triglycerides and cholesterol. Plasma samples will be used for the extraction of brain derived extracellular vesicles. miRNA will be extracted from the Dried Blood Spots and sent for sequencing analysis. Buccal samples will be extracted for DNA and subsequently genotyped while saliva samples will be used to analyze levels of C-Reactive Protein, TNF-alpha, IL-6, IL-8 and IL-1β. Any sample or derivative that is not completely depleted by initial analysis will be retained for future developments or repeats as needed
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Help seeking group: Primary care mental health service providers within the CIUSSS-ODIM catchment area will be the major referral source for this group. Youth and families referred to or self-referring for mental health needs to CLSCs at Dorval-Lachine-LaSalle, CLSC Pierrefonds/Lac-Saint-Louis, Social Paediatrics Clinics and Aire-Ouverte centres throughout the CIUSSS-West Island catchment will be approached by a member of these programmes to assess interest. A screening contact (on site or via telephone) by a member of the research team (who will work on site with clinical teams) will follow to review eligibility criteria. To increase uptake and reduce clinician burden, information leaflets and posters will be made available at the waiting rooms, webpages and social media sites of these youth programmes.
- Non help seeking group: Parents referral pathway: Youth will be recruited through their parents, patients of psychiatric clinics at the CIUSSS-ODIM. Parents will be approached by health professionals. A screening contact by a member of the research team will follow to review eligibility criteria. Other form of recruitment is non-profit organisations serving people living with mental illness, such as the Schizophrenia Society of Quebec as well as primary care practitioners caring for parents satisfying the eligibility criteria. Information leaflets and posters will be made available at the waiting rooms of these clinics and shared with the partner agencies. Social agencies referral pathway: Youth who have contacts with community agencies that provide various forms of social assistance will be recruited through printed and digital advertising. Direct contacts as well as referrals from agency workers and volunteers will be screened by a member of the research team. Physical health based referral pathway: Adv

SUMMARY:
Behavioural Development, Long-term Outcomes and Opportunities to Optimize Youth Mental Health (BLOOM) is a project that aims to overcome age and diagnostic boundaries to generate person-specific longitudinal profiles of mental health in youth aged 9 to 25. The overarching objective is to lay the informational foundation to accurately predict both clinical outcomes and opportunities to optimize health trajectories. This project will recruit youth in need without any mental health diagnosis and follow them annually for 5 years. The present study includes assessment of antecedents, opportunities and outcomes that will establish eligibility for preventive interventions

DETAILED DESCRIPTION:
We propose an accelerated longitudinal study design that allows covering a long developmental period (9 to 25 years) in a short study time (5 years follow-up). Youth and family caregivers will be recruited from various sources and followed-up annually for the first five years. Beyond this 5-year period, further follow-ups will depend on continued study funding and may be either annual or less frequent (e.g. every 3-4 years), and either interview-based or restricted to administrative data. The present study includes assessment of antecedents, opportunities and outcomes that will establish eligibility for preventive interventions; any randomised intervention studies based on this cohort will be based on the outcome for specific REB submissions in the future.

Predicting the onset of DMDs using a set of readily accessible antecedents

We hypothesise that youth who develop DMDs will have higher severity and frequency of antecedents compared to those who do not develop this outcome. We anticipate that a clinically meaningful prediction (i.e., with accuracy 80% or more said to be good or excellent, while less than 60% is deemed not meaningful; many existing predictors perform at 60-80% range9) of DMDs can be made with the set of readily measurable antecedents. We will estimate the strength of antecedent-outcome relationship separately in the two (help-seeking or non help-seeking) subgroups. While we expect variations in the rates of outcomes (help-seeking > non-help seeking), we hypothesise that the relationship between antecedents and DMDs will be similar across the groups with no major drop in the ability to predict outcome in any subgroup (i.e. >60% accuracy in each, below which prediction is unlikely to be of any clinical benefit59).

Relationship between predictive antecedents, resilience and biobehavioural markers

In the consenting subsample, we will assess if the polygenic risk of individual disorders/pathways and summary measures of brain health (age-appropriate structure, chemisty, function) differ between those who develop DMDs and those who do not. We will subsequently test if measures with highest effect size differences, if any, will improve the accuracy (discrimination index) for outcome prediction by at least 10% to assess their suitability for routine clinical implementation.

Of note, we propose this study as a part of a longer program whose first phase will be for 5 years duration. We anticipate following up this cohort for a longer period in phase 2, and embedding clinical trials in the cohort in future (not described here).

ELIGIBILITY:
Inclusion Criteria:

Youth between 9 to 25 years of age at inclusion, who are able to read and understand either French or English, with at least one parent or legal guardian available to consent for those under 18 years of age.

Specific eligibility criteria:

Help-seeking group: At least one help-seeking contact made with a primary care clinical service provider or agency (e.g, paediatric/family physician clinic, CLSC or Aire Ouverte) for a mental health concern (i.e., clinical needs).

Non help-seeking group:

At least one of the birth parents or siblings have received psychiatric care for a diagnosis of DMDs (i.e., family needs) OR Being in contact with community agencies that provide youth-centred social services for food, housing, social discrimination (e.g., racialized youth, LGBTQ2SIA+) (i.e., social needs) OR Having a diagnosed chronic physical illness that is expected to require treatment for >12 months (e.g., diabetes, asthma to name a few) (i.e., physical health needs)

Exclusion Criteria:

* Due to the requirements of assessment procedures, youth who cannot communicate verbally due to known neurological conditions or intellectual disabilities will not be included. Youth who are already diagnosed with one of the DMDs by a physician and currently prescribed a treatment targeting the diagnosed condition (pharmacological or psychotherapeutic interventions), will not be eligible for inclusion.

Importantly, no one will be excluded based on sex, gender, health insurance status, ethnicity, income status, ability to travel or living arrangements. If a participant initially approached through the referral pathways for non help-seeking individuals turns out to have had at least one help-seeking contact for a mental health concern (i.e., clinical needs), the participant will still be included but classified as part of the help-seeking group. We anticipate non help-seeking referrals to satisfy more than one criteria. Their occurrence and distribution will be recorded in detail as part of our assessment procedure.

Ages: 9 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Help-seeking group: Primary care mental health service providers within the CIUSSS-ODIM catchment area will be the major referral source for this group. Youth and families referred to or self-referring for mental health needs to CLSCs at Dorval-Lachine-LaSalle, CLSC Pierrefonds/Lac-Saint-Louis, Social Paediatrics Clinics and Aire-Ouverte centres throughout the CIUSSS-West Island catchment will be approached by a member of these programmes to assess interest. A screening contact (on site or via telephone) by a member of the research team (who will work on site with clinical teams) will follow to review eligibility criteria. To increase uptake and reduce clinician burden, information leaflets and posters will be made available at the waiting rooms, webpages and social media sites of these youth programmes (See the leaflet: Portraying Your Mental Health).
  Non help-seeking group: Parents referral pathway: For this group, youth will be recruited through their parents, who are current
Sampling Method: Non-Probability Sample
Enrollment: 560 (Estimated)
Dates: Start 2024-07-01 (Actual); Primary Completion 2029-07-01 (Estimated); Study Completion 2029-07-01 (Estimated)

PRIMARY OUTCOMES:
Number of new onsets of one of the seven mental illnesses as per DSM-5 criteria | From screening to 5 years of follow-up.
  By applying a detailed diagnostic screen we will be able to capture all emerging mental illnesses as per the existing schedule of classification if present. But our primary outcome of interest (DMDs) is defined as a new onset of illnesses known to involve substantial functional impairment over multiple domains. These are moderate/severe major depressive disorder, bipolar disorder type I or type 2, schizoaffective disorder, schizophrenia, or schizophreniform disorder, anorexia and bulimia nervosa, OCD, moderate/severe ADHD, moderate or severe substance use disorder (SUD) all according to DSM-5 (as per DSM-5 Text Revision, updated September 2023). Notably, while epidemiological data indicates that features of some of these disorders (e.g. ADHD, OCD) begin at ages younger than 9, the mean age of diagnosis continues to be much later in practice.

OTHER OUTCOMES:
Time-to-onset of severe psychopathology based on InterRAI instrument | baseline, 1,2,3,4 and 5 years
  In addition to primary diagnostic outcomes, we assess psychopathology in detail using in-person clinical interviews, speech recordings, self reports and parental reports. The scales used for this purpose are those embedded in the InterRAI child and youth module as well as self-report scales. Time-to-onset for the first supra-threshold symptom will be measured in each subject (reported in months since first observation)

CONTACTS AND LOCATIONS:
Locations (1):
- Centre intégré universitaire de santé et de services sociaux (CIUSSS) de l'Ouest-de-l'Île-de-Montréal, Montreal, Quebec, Canada